CLINICAL TRIAL: NCT07252609
Title: Effects of Oral Sodium Butyrate Supplementation on Body Weight Reduction in Overweight/Obese Individuals With and Without Type 2 Diabetes
Acronym: ButRed
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Giuseppina Costabile, Senior Researcher, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 44/2024
Record Dates: First submitted 2025-11-17; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Obesity; Type 2 Diabetes
Keywords: Butyrate; body weight; obesity; type 2 diabetes; butyrate supplementation; glucose control; lipid metabolism
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Body Weight | interventions — Butyric Acid

STUDY DESIGN:
Intervention Model Description: The experimental study will be conducted according to a randomized parallel-group design, involving 46 obese individuals, with and without type 2 diabetes. The experimental phase will be preceded by a 3-week observation period (run-in), during which participants will stabilize their habitual diet. At the end of this period, participants will be randomly assigned to one of two 12-week treatments:
  1. oral supplementation with sodium butyrate (NaBut) + hypocaloric diet, or
  2. oral supplementation with placebo + hypocaloric diet.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Sodium Butyrate Supplementation (NaBut) (Experimental): Participants receive oral sodium butyrate (NaBut) in combination with a moderately hypocaloric diet. Sodium butyrate is administered in tablet form (Butir Bioma®, UNIFARCO S.p.A.), with each tablet containing 625 mg of sodium butyrate. Participants take one tablet three times daily-at breakfast, lunch, and dinner-for a total daily dose of 1,875 mg.
  Interventions: Dietary Supplement: Sodium Butyrate (NaBut)
- Placebo (Placebo Comparator): Participants receive placebo tablets in combination with the same moderately hypocaloric diet as the experimental group (NaBut arm).
  The placebo tablets are identical in appearance, weight, shape, color, and taste to the sodium butyrate tablets but do not contain the active ingredient (sodium butyrate).
  Participants take one placebo tablet three times daily-at breakfast, lunch, and dinner-for a total of three tablets per day.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Sodium Butyrate (NaBut) — Participants receive oral sodium butyrate (NaBut) in combination with a moderately hypocaloric diet for 12 weeks.
  Sodium butyrate is administered as 625 mg tablets (Butir Bioma®, UNIFARCO S.p.A.), taken three times daily with meals (breakfast, lunch, and dinner), for a total daily dose of 1,875 mg.
  The hypocaloric diet is individualized based on basal metabolic rate (measured by indirect calorimetry) and physical activity level, with a 300-500 kcal/day energy reduction.
  Arms: Oral Sodium Butyrate Supplementation (NaBut)
Dietary Supplement: Placebo — Participants receive placebo tablets identical in appearance, weight, shape, color, smell, and taste to the sodium butyrate tablets but without the active ingredient, combined with the same moderately hypocaloric diet as the experimental group.
  Tablets are taken three times daily with meals (breakfast, lunch, and dinner), for a total of three tablets per day.
  The hypocaloric diet follows the same composition and energy restriction as described for the sodium butyrate intervention.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial (randomized controlled trial with parallel group design) is to evaluate the effects of oral sodium butyrate supplementation for 12 weeks, compared with placebo, in addition to a moderately hypocaloric diet, on body weight, body composition, glucose metabolism, and lipid metabolism in overweight or obese individuals with and without type 2 diabetes.

The main questions this study aims to answer are:

* Does oral sodium butyrate improve body weight reduction and body composition compared with placebo?
* Does it improve glucose and lipid metabolism in participants with and without type 2 diabetes?

The study includes 46 men and women aged 30-70 years, with overweight or obesity (BMI 25-39.9 kg/m²) and HbA1c ≤ 7.0%. Participants are randomly assigned to receive either oral sodium butyrate or placebo, both combined with a moderately hypocaloric diet for 12 weeks.

Participants:

* Take sodium butyrate tablets (625 mg three times daily; total 1,875 mg/day) or placebo tablets with meals
* Follow a personalized, balanced hypocaloric diet monitored by a dietitian
* Attend clinic visits every two weeks for anthropometric measurements and dietary adherence checks
* Complete a 7-day food diary and a gastrointestinal symptom questionnaire (PAGI-SYM)
* Undergo fasting blood tests, body composition analysis (bioelectrical impedance), and continuous glucose monitoring (CGM) at baseline and after 12 weeks

ELIGIBILITY:
Inclusion Criteria:

* Men and women with overweight or obesity (Body Mass Index [BMI] between 25.0 and 39.9 kg/m²), with or without type 2 diabetes Age between 30 and 70 years HbA1c ≤ 7.5%

Exclusion Criteria:

* Cardiovascular events (myocardial infarction and/or stroke) within the previous 6 months
* Renal insufficiency (serum creatinine > 1.5 mg/dL) or hepatic impairment (ALT or AST levels more than twice the upper limit of normal)
* Anemia (hemoglobin < 12 g/dL)
* Insulin therapy or use of antihyperglycemic drugs other than metformin
* Use of antibiotics, probiotics, or prebiotics within the previous 3 months
* Habitual intense physical activity
* Pregnancy or breastfeeding

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2024-11-13 (Actual); Primary Completion 2025-08-08 (Actual); Study Completion 2025-08-08 (Actual)

PRIMARY OUTCOMES:
Reduction in Body Weight After 12 Weeks of Oral Sodium Butyrate Supplementation Compared With Placebo | baseline and 12 weeks
  Body weight is measured at baseline and after 12 weeks of treatment. The primary outcome is the reduction in body weight (kg) from baseline to week 12 between the sodium butyrate and placebo groups.

SECONDARY OUTCOMES:
Change in Body Composition (Fat Mass, Lean Mass, and Fat-Free Mass) | baseline and 12 weeks
  Body composition is assessed by bioelectrical impedance analysis (BIA) at baseline and after 12 weeks to evaluate changes in fat mass, lean mass, and fat-free mass between groups.
Changes in Continuous Glucose Monitoring (CGM) Parameters | baseline and 12 weeks
  Continuous glucose monitoring (CGM) is performed for 7 days at baseline and at the end of treatment to evaluate mean glucose levels, variability, and time-in-range between groups.
Changes in Fasting Glucose | Baseline and 12 weeks
  Fasting plasma glucose is assessed at baseline and at week 12 by immunoenzymatic assay; results are reported in mg/dl
Changes in fasting insulin | Baseline and 12 weeks
  Fasting plasma insulin is assessed at baseline and at week 12 by ELISA method and expressed in µU/ml
Changes in glycated hemoglobin (HbA1c) | Baseline and 12 weeks
  Glycated hemoglobin (HbA1c) was measured at baseline and after 12 weeks in fasting whole-blood samples by high-performance liquid chromatography (HPLC) and was expressed as mmol/mol and %.
Changes in serum lipids | Baseline and 12 weeks
  Fasting serum triglycerides, total cholesterol and HDL cholesterol are evaluated at baseline and after 12 weeks using immunoenzymatic methods and all expressed in mg/dL
Changes in Short-Chain Fatty Acids (SCFA) | Baseline and 12 weeks
  Serum concentrations of short-chain fatty acids (acetate, propionate, butyrate) are measured at baseline and after 12 weeks.
  SCFA levels are assessed as metabolic markers of gut microbial activity and host metabolic response to sodium butyrate supplementation. They were quantified by gas chromatography with flame ionization detection (GC/FID) and expressed in μmol/L
Changes in Intestinal Permeability Markers_Zonulin | Baseline and 12 weeks
  Fasting serum zonulin, as a biomarker of intestinal permeability, is measured at baseline and after 12 weeks by ELISA and expressed in ng/mL
Changes in Intestinal Permeability Markers_LPS | Baseline and 12 weeks
  Fasting serum lipopolysaccharide (LPS), a biomarker of intestinal permeability, is measured at baseline and after 12 weeks by ELISA and expressed in pg/mL
Changes in Inflammatory Markers_hsCRP | Baseline and 12 weeks
  Serum high-sensitivity C-reactive protein (hs-CRP) concentrations are measured at baseline and after 12 weeks using immunoturbidimetric methods and expressed in mg/dL
Changes in Gut Microbiota Composition | baseline and 12 weeks
  Fecal samples are collected at baseline and after 12 weeks to evaluate the effects of sodium butyrate on gut microbiota composition, compared to placebo. Microbial community structure is analyzed using 16S rRNA gene sequencing and shotgun metagenomic techniques to assess taxonomic and functional changes
Changes in Inflammatory Markers_TNFalfa_IL-6 | Baseline and 12 weeks
  Serum tumor necrosis factor-alpha (TNF-α) and interleukin-6 (IL-6) concentrations are measured at baseline and after 12 weeks using ELISA and are expressed in pg/mL

CONTACTS AND LOCATIONS:
Overall Officials: Lutgarda Bozzetto, Full Professor, Principal Investigator — Federico II University
Locations (1):
- Federico II University, Napoli, Italy

IPD SHARING:
Plan to Share IPD: No
no secure institutional infrastructure is currently available to support anonymized data sharing